CLINICAL TRIAL: NCT02693483
Title: Preoperative Vaginal Cleansing With Povidone Iodine and the Risk of Post Cesarean Endometritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: povidone iodine
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Infection; Cesarean Section
MeSH Terms: conditions — Infections | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- povidone iodine (Active Comparator): 153 cases undergoing cesarean sections will have preoperative vaginal cleansing with 10% povidone iodine
  Interventions: Drug: 10% povidone iodine
- no vaginal cleansing (No Intervention): 153 cases undergoing cesarean sections

INTERVENTIONS:
Drug: 10% povidone iodine — Vaginal cleansing will be done with 3 gauze pieces soaked with 10% povidone iodine in a sterilized bowl and the scrub will be done from the vaginal apex to introitus with attention to the anterior, posterior and lateral vaginal wall
  Other Names: betadine
  Arms: povidone iodine

SUMMARY:
Preoperative vaginal cleansing with povidone iodine and the risk of post cesarean endometritis.

DETAILED DESCRIPTION:
Study Population:

Women undergoing cesarean sections will be enrolled in this study after obtaining verbal consent as there are no extra interventional measures that will be undertaken in the study apart from routine investigations and procedures done during cesarean sections, being already approved in signed consent to undergo treatment.

The nature and aim of the work will be fully discussed to all women who will agree to participate in the study. Verbal consent will be obtained from all patients enrolled in the study which is approved by the local ethical committee.

Preoperative evaluation of patients included:

1. Medical history taking including:

   * Personal (name, age)
   * Complaint (in patient word)
   * Present history
   * Medical history (Diabetes mellitus, Hypertension)
   * Past history (any surgeries)
   * Family history
2. Physical examination including vital data (blood pressure,pulse, temperature)
3. Routine hematologic laboratory tests including complete blood picture & random blood sugar.
4. The surgical site will be assessed at least once before cesarean section if the participant presented to emergency department with findings concerning for surgical-site infection.
5. Indication for cesarean section.
6. Duration of ruptured membranes if found.
7. Risk of infection including Diabetes mellitus, immuno-compromised, rupture of membranes and corticosteroid therapy.

Steps:

Patients In the study group (povidone iodine group) patients will be prepared with vaginal cleansing with povidone-iodine along with the usual abdominal scrub. Vaginal cleansing will be done with 3 gauze pieces soaked with 10% povidone iodine in a sterilized bowl and the scrub will be done from the vaginal apex to introitus with attention to the anterior, posterior and lateral vaginal wall. After vaginal cleansing the gloves will be changed to perform the abdominal scrub.

Patients in the control group (no vaginal cleansing group) will not have any vaginal wash (even tap water will not be used).

In both groups, patients will receive preoperative per protocol prophylactic I.V. antibiotics (third generation cephalosporin ) before skin incision.

Operative technique:

During this study all cases will be subjected to exclusion and inclusion criteria. Any risk of infection will be assessed including rupture of membranes, Diabetes mellitus, immune-compromised and corticosteroid therapy….etc. Cesarean section will be performed with estimation of operative duration in time and mean operative blood loss.

Post operative care:

Follow up for temperature of 38°C and greater during first 24 hours of surgery and endometritis will be diagnosed by fever 38.4°C and greater with any of the following (uterine tenderness ,foul smelling lochia or positive C-reactive protein).

Mean hospital stay in days will be determined. N.B: Culture of the upper genital tract are virtually impossible to obtain without contaminating the specimen by the microorganisms in the vagina. Therefore, they rarely add significant information that enhances clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-40 years of age who will undergo cesarean deliveries.
2. Able to communicate well with the investigator & to comply with the requirements of the entire study.
3. Verbal consent obtained from subject and husband / witness before undergoing the study entry (with the understanding that consent may be withdrawn by the patient at any time without prejudice).

Exclusion Criteria:

1. Patients with allergy to iodine containing solutions.
2. Patients with ante-partum hemorrhage.
3. Patients with ruptured membranes.
4. Patients with any known disease that increases the risk of infection e.g. immunocompromized, those receiving steroids ...etc.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 306 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with post cesarean endometritis | 48 hours
  Number of Subjects with post cesarean endometritis as diagnosed by fever 38.4°C and greater in first 48 hours after cesarean section with any of the following (uterine tenderness, foul smelling lochia or positive C-reactive protein)

SECONDARY OUTCOMES:
Number of Subjects with allergic reaction to povidone iodine | 48 hours
  Number of Subjects with allergic reaction to povidone iodine

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895